CLINICAL TRIAL: NCT07258316
Title: Comparative Effects of High-Intensity Interval Training in Pre and Postmenopausal Women With Type II Diabetes Mellitus
Brief Title: High Intensity Interval Training in Pre and Postmenopausal Women With Type II Diabetes.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mushafaeen Rizwan
Record Dates: First submitted 2025-08-24; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Postmenopausal Symptoms
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — High-Intensity Interval Training; Warm-Up Exercise

STUDY DESIGN:
Intervention Model Description: There will be comparison between the two groups, experimental and control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training group (Experimental): The group will receive 8 weeks of High Intensity Interval Training (27 sessions, 3/week, 60-90 minutes). Progresssion for 1-4 weeks will of Workout Interval : Rest Interval will be 30 sec : 30 sec of each exercise and from week 5-8 the progression will be 30 sec : 15 sec. Both Warm-up and Cool down exercises will be of 10-15 minutes.
  Interventions: Other: High Intensity Interval Training (warm up, Mat exercises,cycling,HIIT exercises,cool down)
- Control group (Active Comparator): This group will receive Resistance Exercises with alternate days 3 times per week for 8 weeks and total sessions will be 27. Both warmup and cool down will be of 10-15 minutes and progression will be increased gradually. This group will include different Resistance Exercises and the time duration will be 60-90 minutes
  Interventions: Other: Control (warm up, Mat exercises,cycling,Resistance exercises,cool down)

INTERVENTIONS:
Other: High Intensity Interval Training (warm up, Mat exercises,cycling,HIIT exercises,cool down) — This will include 8 weeks of plan with total 27 sessions 3 times a week and each session will include warm up exercises ( Treadmill (Incline and Reverse), Mat Exercises (Cobra, Cat/camel stretches, Superman, Aeroplane and Skydiving exercises)and Cycling (Seated and un-supported). this will be of 10-15 minutes. Then HIIT exercises which includes High knees, Push ups, Russian crunches, Battle ropes, Weighted squats, Planks, Seated rows and Jumping jacks. Then cool- down exercises will be of 10-15 minutes and this will includes Full body Stretches (Quadriceps, Hamstrings, Piriformis, Calfs, Biceps, Triceps, Rhomboids, IT band, Trapezius, and Chest Stretches), whole exercise plan will take 60-90 minutes.
  Arms: High Intensity Interval Training group
Other: Control (warm up, Mat exercises,cycling,Resistance exercises,cool down) — This group will includes also recieve 8 weeks of exercises plan for 3/week warmup exercises same as the experimental group such as Treadmill (Incline and Reverse), Mat Exercises (Cobra, Cat/camel stretches, Superman, Aeroplane and Skydiving exercises)and Cycling (Seated and un-supported) forv about 10-15 miutes Resistance Exercises like (LAT Pull down, Leg Curls, Leg Extension, Hips Adductor/ Abductors, Seated Rowing, Rear deltoid machine). the progression will be increased gradually. Cool down exercises includes full body streching and the whole session will be of 60-90 minutes
  Arms: Control group

SUMMARY:
Diabetes Mellitus (DM), a chronic metabolic disease-causing chronic hyperglycemia. Globally more than 90% cases are of type II diabetes mellitus (T2DM). Around 537 million adults worldwide had diabetes but according to data from Pakistan, female sufferers are marginally higher (26.4%) as compared to men (25.1%). The main causes of DM II are genetic predispositions, including consanguinity, dietary changes, urbanization and sedentary lifestyles. It is reported that postmenopausal status is linked to worsened glycemic control, increased visceral adiposity and and inflammation, and women before menopause generally have improved lipid metabolism and insulin sensitivity. HIIT provides powerful and time-efficient benefits by alternating high-intensity workouts (85-95% HR_Max) with recovery.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM), is linked to impaired protein, lipid and carbohydrate metabolism, as well as impaired insulin secretion or its reduced sensitivity and this number will increase to almost 643 million by 2030 and 783 million by 2045. As estimated by the International Diabetes Federation (2021), the burden of DM type II is especially severe in Pakistan, where 33 million adults are affected by it, ranking Pakistan at number three globally. A study published in January 2025 in BMC Public Health found that the DALY burden of type 2 diabetes in Asian women was approximately 7,122 per 100,000, with behavioral risk factors (air pollution, fasting plasma glucose, and dietary risks) playing a significant role. The Study of Women's Health across the Nation (SWAN) cohort showed that Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) levels rose steadily during menopause this means that insulin resistance gets a lot worse for women during menopause. While another study reported that postmenopausal women have comparatively increased Low Density Lipo-protein (LDL) cholesterol, triglycerides, decreased high-density lipoprotein (HDL) cholesterol, increased C-Reactive Protein (CRP) and Interleukin-6 (IL-6), the markers of cardio-metabolic risk, as compared to premenopausal women. As estradiol deficiency is linked to decreased adiponectin and increased leptin, these hormonal changes also upset the balance of adipokines, exacerbating insulin resistance and inflammatory signaling pathways. After age 45, the odds ratio (OR) of getting T2DM was about 0.13, and the risks stopped rising after age 50-55. The key to managing type 2 diabetes is physical activity. Insulin sensitivity, systemic inflammation, fasting glucose, and HbA1c are all improved by conventional aerobic exercise. High-intensity interval training (HIIT) and other interventions meant to improve insulin sensitivity and inflammatory status. HIIT improves mitochondrial function, decreases inflammation, changes the distribution of body fat, and increases muscle glucose uptake to help manage type 2 diabetes in premenopausal and postmenopausal women. HIIT therefore enhances insulin sensitivity and glycemic control. According to meta-analyses, adults with type 2 diabetes who receive 8-12 weeks of HIIT experience significant decreases in their HbA1c (0.3-0.8%), fasting insulin (~20-30%), and CRP (~15-25%). In another study HIIT protocol were applied on the PCOS women with hormonal imbalances and metabolic issues Running at 100-110% of maximum aerobic velocity (MAV) was part of the training regimen, which was divided into 4-6 sets of 4 laps. For eight weeks, participants trained three times a week. The goal of this intense training program was to improve aerobic capacity and performance. Diabetes is prevalent worldwide; postmenopausal women are more vulnerable because of metabolic and hormonal changes. Previous studies have not much inquired the effect of glycemic control in varying menopausal status, although effectiveness of HIIT is proven for improving in insulin sensitivity and CRP in women and is considered a promising modality, but there is need to determine its effectiveness across women of varied menopausal status with T2DM. The aim of the study is to evaluate the effects of HIIT on glycemic control, Inflammatory markers, and Insulin sensitivity in pre versus postmenopausal women with T2DM and to support culturally appropriate menopause-sensitive exercise recommendations for women with T2DM.High-Intensity Interval Training (HIIT) provides a quick, non-pharmacological method to enhance insulin sensitivity, blood sugar regulation, body composition, and heart health, , this study intends to investigate how HIIT can specifically help manage blood sugar problems associated with hormonal changes associated with menopause.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 40-65 years with physician-diagnosed T2DM.
* Premenopausal (regular menstruation) or postmenopausal (≥12 months amenorrhea) (self-reported).
* Participants who have not engaged in any structured exercise sessions or gym workouts in the past six months.
* Willing to follow supervised HIIT protocol and provide informed consent.

Exclusion Criteria:

* Cardiovascular, orthopedic, or endocrine conditions contraindicating exercise.
* Current use of insulin or hormone replacement therapy.
* Participation in structured exercise programs in the past 6 months.
* Cognitive impairment or psychiatric illness

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline and 8 weeks
  For monitoring long-term glycemic control, the average blood glucose over the past 2-3 months.
  its values range from Normal: < 5.7%, Prediabetes: 5.7% - 6.4%, Diabetes: ≥ 6.5%
Fasting Blood Glucose | Baseline and 8 weeks
  For Assessing short-term blood sugar control, used for onitoring glucose levels in metabolic disorders and Screening for insulin resistance or hypoglycemia..
  Normal: 70 - 99 mg/dL (3.9 - 5.5 mmol/L), Prediabetes: 100 - 125 mg/dL (5.6 - 6.9 mmol/L), Diabetes: ≥ 126 mg/dL (≥ 7.0 mmol/L)
Fasting Insulin | Baseline and 8 week
  Evaluating insulin resistance and sensitivity also use to monitoring and managing diabetes).
  Normal: 2 - 20 µU/mL
Basic Lipid Profile testing including total cholesterol, Low-Density Lipoprotein-Cholesterol,High-Density Lipoprotein-Cholesterol and Triglycerides. | Baseline and 8 week
  these are validated blood tests for diagnosing dyslipidemia. A lipid profile's normal ranges, in mg/dL, are: Total Cholesterol: < 200, LDL (Bad) Cholesterol: < 100 (or < 70 for those with diabetes), HDL (Good) Cholesterol: > 60, and Triglycerides: < 150
CRP | Baseline and 8 week
  for Detecting and monitoring inflammation in the body) Normal: < 10 mg/L Elevated: > 10 mg/L
QUICKI (Quantitative Insulin Sensitivity Check Index) | Baseline and 8 week
  Normal value ≥ 0.33.
  * Estimating insulin sensitivity (higher = better sensitivity)
  * An alternative to HOMA-IR, especially in research settings.
HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) | Baseline and 8 week
  Normal value < 2
  * Estimating insulin resistance (higher = more resistance)
  * Early detection of metabolic syndrome, prediabetes, or type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PhD, Principal Investigator — Riphah Itnernational University, Islamabad Pakistan
Locations (1):
- Ginnastic Health Centre, Islamabad, Islamabad, Islamabad Capital Territory, Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Motahari-Tabari N, Ahmad Shirvani M, Shirzad-E-Ahoodashty M, Yousefi-Abdolmaleki E, Teimourzadeh M. The effect of 8 weeks aerobic exercise on insulin resistance in type 2 diabetes: a randomized clinical trial. Glob J Health Sci. 2014 Aug 14;7(1):115-21. doi: 10.5539/gjhs.v7n1p115. PMID 25560330
- [Background] Mandrup CM, Egelund J, Nyberg M, Enevoldsen LH, Kjaer A, Clemmensen AE, Christensen AN, Suetta C, Frikke-Schmidt R, Steenberg DE, Wojtaszewski JFP, Hellsten Y, Stallknecht BM. Effects of menopause and high-intensity training on insulin sensitivity and muscle metabolism. Menopause. 2018 Feb;25(2):165-175. doi: 10.1097/GME.0000000000000981. PMID 28953212
- [Background] Cybulska AM, Schneider-Matyka D, Wieder-Huszla S, Panczyk M, Jurczak A, Grochans E. Diagnostic markers of insulin resistance to discriminate between prediabetes and diabetes in menopausal women. Eur Rev Med Pharmacol Sci. 2023 Mar;27(6):2453-2468. doi: 10.26355/eurrev_202303_31779. PMID 37013763